CLINICAL TRIAL: NCT00782457
Title: Prospective Randomised Study Comparing Laparoscopic Versus Open Surgery in Patients With Rectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Universitario Virgen de la Arrixaca (Other)
Responsible Party: Juan Lujan, HUV Arrixaca
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D-08-00770
Record Dates: First submitted 2008-10-29; First posted 2008-10-31 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2008-10

CONDITIONS: RECTAL CANCER
MeSH Terms: conditions — Rectal Neoplasms

ARMS (2):
- OPEN SURGERY (Active Comparator)
  Interventions: Procedure: RECTAL CANCER RESECTION
- LAPAROSCOPIC SURGERY (Experimental)
  Interventions: Procedure: RECTAL CANCER RESECTION

INTERVENTIONS:
Procedure: RECTAL CANCER RESECTION

SUMMARY:
The aim of this study is to compare laparoscopic versus open approach on the surgical treatment of mid and low-lying rectal cancer, both performed by the same surgical team with experience in open colorectal surgery and advanced laparoscopic surgery, assessing preoperative and anatomopathological results and long-term outcome.

ELIGIBILITY:
Inclusion Criteria:

* Mid- and low-lying rectal cancer (between 0 and 11 cm from the anal margin)
* Histology of adenocarcinoma

Exclusion Criteria:

* Locally advanced disease (T4)
* Emergency surgery
* Rectal cancer over familial colic polyposis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2002-01; Primary Completion 2007-02 (Actual); Study Completion 2010-12

PRIMARY OUTCOMES:
Lymph nodes isolated, circumferential margin involved, rate of complications and length of stay | 1 month

REFERENCES:
- [Derived] Lujan J, Valero G, Hernandez Q, Sanchez A, Frutos MD, Parrilla P. Randomized clinical trial comparing laparoscopic and open surgery in patients with rectal cancer. Br J Surg. 2009 Sep;96(9):982-9. doi: 10.1002/bjs.6662. PMID 19644973